CLINICAL TRIAL: NCT02370069
Title: The Effect of Previous Pneumococcal Immunization on the Immune Response of Adult Patients With Severe Chronic Kidney Disease to Prevnar 13
Brief Title: The Effect of Previous Pneumococcal Immunization on the Immune Response of Patients With Severe CKD to Prevnar 13
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Marina Ulanova, Associate Professor, Division of Medical Sciences, Lakehead University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RP-232-08262014
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Previous immunization with PPV23 (Active Comparator): Participants who have received a previous vaccination with 1 or more dose of PPV23 at least 12 months previously will receive one dose of 0.5 mL Prevnar 13 study vaccine.
  Interventions: Biological: Prevnar 13
- Naive to PPV23 (Active Comparator): Participants who have never received a previous vaccination with PPV23 will receive one dose of 0.5 mL Prevnar 13 study vaccine.
  Interventions: Biological: Prevnar 13

INTERVENTIONS:
Biological: Prevnar 13 — One dose of 0.5 mL Prevnar 13 injected intramuscularly into the deltoid muscle on Day 0.

SUMMARY:
Patients with severe chronic kidney disease (CKD) are at a great risk for infection due to their immune system being suppressed. Pneumococcal infection is particularly common and often results in death due to inflammation of lung (pneumonia) or the whole body (sepsis). This infection can be prevented using vaccines which help build protective immunity. The currently recommended pneumococcal vaccine (Pneumovax), however, is often inefficient in this group of patients. There is thus an urgent need to improve the existing vaccination policy.

The goal of this research is to optimize pneumococcal vaccination of patients with severe CKD. Many patients suffering from CKD have already been vaccinated with Pneumovax. Because this vaccine has low immunogenicity in immunocompromised individuals, they may still develop infection. A new vaccine, Prevnar13, has superior immunogenicity and has been recently approved for immunization. There is, however, no specific policy regarding immunization of adult CKD patients, and it is furthermore unknown whether previous Pneumovax immunization negatively affects immune response to Prevnar13.

In order to test whether previous immunization with Pneumovax affects the immune response of severe CKD patients to Prevnar 13, the investigators will immunize two groups of adult stage 4 and 5 CKD patients with one dose of Prevnar 13 and will assess their initial immunological response, its longevity, and vaccine safety. The first group will consist of patients who had been previously immunized with Pneumovax, and the second group will include participants with no history of pneumococcal vaccination.

Antibody levels and opsonophagocytic activity (OPA) will be quantified. The longevity of the immune response will be assessed. As a secondary objective, the immune response will be analyzed in the context of demographic and clinical characteristics of the vaccinated participants.

DETAILED DESCRIPTION:
Adult patients with severe chronic kidney disease (CKD) are immunocompromised and known to have an increased risk of pneumococcal infection. To prevent the infection, immunization with pneumococcal polysaccharide vaccine (PPV23) is currently recommended in Canada; however, the vaccine effect in these patients is suboptimal because of their immune dysfunction. The second-generation pneumococcal vaccines (polysaccharide-protein conjugate) have superior immunogenicity in some immunocompromised adult individuals. In Canada, Prevnar 13 has recently been recommended by the NACI for certain categories of immunocompromised adults, such as HSCT recipients and HIV-positive patients. However, the NACI has concluded that there is currently insufficient evidence to recommend the use of Prevnar 13 in patients with chronic kidney disease. No published data on the use of pneumococcal conjugate vaccines in adults with CKD are available. Moreover, it is unknown whether a previous immunization with PPV23 may have a negative effect on the immune response to Prevnar 13 in these patients. Such a possibility exists due to the memory B-cells' depletion following immunization with pure polysaccharide antigens. In this case, additional doses of Prevnar 13 may be required to achieve the optimal protection. The conjugate vaccine will then expand the B-cell pool available to respond to subsequent antigen challenge. To test whether previous immunization with PPV23 affects the immune response of severe CKD patients to Prevnar 13, we will immunize two groups of adult stage 4 and 5 CKD patients attending the Thunder Bay Regional Health Sciences Centre with one dose of Prevnar 13 and will assess their initial immunological response, its longevity, and vaccine safety. The first group will consist of patients who had been immunized with PPV23 more than one year prior to the enrollment in this study and the second group will include patients without history of pneumococcal vaccination. Fold increase in antibody levels and OPA, as well as longevity of the immune response over a one-year period will be assessed as the surrogate for protection against pneumococcal infection. The immune response will be analyzed in the context of demographic and clinical characteristics of the vaccinated patients. All infectious episodes in the study participants will be recorded throughout one year of observation. We will also record all vaccine adverse effects following immunization and compare their frequency and severity between the two groups. The anticipated results of this trial will provide essential evidence to justify the use of Prevnar 13 for immunization of adult CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 18 years of age or older at the time of the vaccination
* Severe chronic kidney disease (Stage 4 and 5)

Exclusion Criteria:

* immunization with PPV23 within the last year
* any confirmed or suspected immunodeficiency condition, including human immunodeficiency virus (HIV) infection, haematological malignancy, or a congenital immunodeficiency
* history of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* history of allergic disease likely to be stimulated by the vaccination
* history or records of immunosuppressive therapy (with the exception of topical corticosteroids) for more than 14 days and within 6 months of vaccination
* history or evidence of administration of immunoglobulins and/or any blood products during the study period or within the three months preceding the study vaccine
* use of any other investigational or non-registered drug or vaccine during the study period or within 30 days preceding the study vaccine
* administration of a vaccine during the period starting one month before the dose of vaccine and ending one month after
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
immunogenicity (Fold increase in serotype-specific antibody levels 28 days post-immunization as compared to baseline) | 0 days, 28 days
  Fold increase in serotype-specific antibody levels 28 days post-immunization as compared to baseline
immunogenicity (Increase in OPA titres 28 days post-immunization) | 28 days
  Increase in OPA titres 28 days post-immunization

SECONDARY OUTCOMES:
Longevity of the immune response (Persistence of antibody one year post-immunization) | 365 days
  Persistence of antibody one year post-immunization
Longevity of the immune response (Persistence of OPA titres one year post-immunization) | 365 days
  Persistence of OPA titres one year post-immunization
Clinical effect (Number of all infectious episodes during one year post-immunization) | 365 days
  Number of all infectious episodes during one year post-immunization

CONTACTS AND LOCATIONS:
Overall Officials: Marina Ulanova, MD, PhD, Principal Investigator — Lakehead University
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulanova M, Huska B, Desbiens A, Gaultier GN, Domonkos V, McCready WG. Immunogenicity and safety of the 13-valent pneumococcal conjugate vaccine in 23-valent pneumococcal polysaccharide vaccine-naive and previously immunized adult patients with severe chronic kidney disease. Vaccine. 2021 Jan 22;39(4):699-710. doi: 10.1016/j.vaccine.2020.12.035. Epub 2020 Dec 24. PMID 33358702
- [Derived] Ulanova M, Huska B, Dubois S, McCready W. Opsonophagocytic activity against Streptococcus pneumoniae in Indigenous and non-Indigenous patients with severe chronic kidney disease immunized with 13-valent pneumococcal conjugate vaccine. Vaccine. 2022 Jul 30;40(32):4594-4602. doi: 10.1016/j.vaccine.2022.06.042. Epub 2022 Jun 21. PMID 35738971
- [Derived] Gaultier GN, McCready W, Ulanova M. The effect of pneumococcal immunization on total and antigen-specific B cells in patients with severe chronic kidney disease. BMC Immunol. 2019 Nov 12;20(1):41. doi: 10.1186/s12865-019-0325-9. PMID 31718534